CLINICAL TRIAL: NCT03007706
Title: Role of Skin Cleansing and Prophylactic Antibiotic in Preventing Infectious Morbidity After Cesarean Section Delivery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Raghda Gamal Mohamed (Other)
Responsible Party: Sponsor-Investigator, Raghda Gamal Mohamed, Minia university, Minia Maternity University Hospital
Organization: Minia Maternity University Hospital (Other)
Other Study IDs: MiniaMUH
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Postpartum Infectious Morbidity in Cesarean Section Delivery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks

INTERVENTIONS:
Procedure: Women undergo cesarean section delivery

SUMMARY:
This study aims to determine the effectiveness of skin cleansing and prophylactic antibiotics given to women undergoing a cesarean section for reducing the incidence of postpartum infectious morbidity and to assess potential maternal adverse effects and any impact on the infant.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing cesarean delivery, both elective and non-elective.
2. Rupture of membranes and labor contractions will be allowed.

Exclusion Criteria:

1. Unknown outcome from the patient.
2. Refusing to participate in the study from the admission conse
3. Allergy to antibiotics.
4. Any visible infection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women undergo cesarean section delivery whether elective or emergency
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
role of skin cleansing and prophylactic antibiotics given to women undergoing a cesarean section for reducing the incidence of postpartum infectious morbidity | 2 weeks following cesarean section